CLINICAL TRIAL: NCT00850044
Title: A Double-Blind, Randomized, Placebo-Controlled, Nonfasting Study in Healthy Adults to Evaluate the Safety, Tolerability, and Pharmacokinetic Profiles of Single Doses of ABT-450 With and Without Ritonavir
Brief Title: Safety, Tolerability and PK Study of Single Doses of ABT-450 With and Without Ritonavir to Treat Hepatitis C Virus (HCV) Genotype 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Adebayo Lawal, M.D./Medical Director, Abbott
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: M10-749
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2010-09

CONDITIONS: HCV Infection
Keywords: FIH; SAD
MeSH Terms: conditions — Hepatitis C | interventions — paritaprevir; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): ABT-450
  Interventions: Drug: ABT-450
- 2 (Placebo Comparator): Placebo for ABT-450
  Interventions: Drug: placebo for ABT-450
- 3 (Active Comparator): ABT-450/ritonavir
  Interventions: Drug: ABT-450; Drug: ritonavir
- 4 (Placebo Comparator): Placebo for ABT-450/placebo for ritonavir
  Interventions: Drug: placebo for ABT-450; Drug: Placebo for ritonavir

INTERVENTIONS:
Drug: ABT-450 — capsules,QD, one dose, see Arm Descriptions for more information
  Arms: 1; 3
Drug: ritonavir — capsules, QD, one dose, escalating doses, see Arm Descriptions for more information
  Other Names: ABT-538; Norvir
  Arms: 3
Drug: placebo for ABT-450 — capsules, QD, one dose
  Other Names: placebo
  Arms: 2; 4
Drug: Placebo for ritonavir — capsules, QD, one dose
  Other Names: placebo
  Arms: 4

SUMMARY:
The purpose of this study is to determine the pharmacokinetic and safety profiles of an experimental HCV protease inhibitor with and without ritonavir in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* overall healthy subjects
* non-childbearing potential females included

Exclusion Criteria:

* history of significant sensitivity to any drug
* positive test for HAV IgM, HBsAg, anti-HCV Ab or anti-HIV Ab
* history of gastrointestinal issues or procedures
* history of seizures, diabetes or cancer (except basal cell carcinoma)
* clinically significant cardiovascular, respiratory (except mild asthma), renal, gastrointestinal, hematologic, neurologic, thyroid, or any uncontrolled medical illness or psychiatric disorder
* use of tobacco or nicotine-containing products with the 6-month period prior to study drug administration
* donation or loss of 550 mL or more blood volume or receipt of a transfusion of any blood product within 8 weeks prior to study drug administration
* abnormal screening laboratory results that are considered clinically significant by the investigator
* current enrollment in another clinical study
* previous enrollment in this study
* recent (6-month) history of drug/alcohol abuse that could preclude adherence to the protocol
* pregnant or breastfeeding female
* requirement for any OTC and/or prescription medication, vitamins and/or herbal supplements on a regular basis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (blood draws, pre- and post-dose) | 4 days
Safety and Tolerability (ECGs, AEs, vitals, physical exams, routine labs) | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Adebayo A Lawal, MD, Study Director — Abbott
Locations (1):
- Site Reference ID/Investigator# 15981, Waukegan, Illinois, United States

REFERENCES:
- [Result] Menon RM, Klein CE, Podsadecki TJ, Chiu YL, Dutta S, Awni WM. Pharmacokinetics and tolerability of paritaprevir, a direct acting antiviral agent for hepatitis C virus treatment, with and without ritonavir in healthy volunteers. Br J Clin Pharmacol. 2016 May;81(5):929-40. doi: 10.1111/bcp.12873. Epub 2016 Feb 24. PMID 26710243